CLINICAL TRIAL: NCT03606447
Title: An Open Label, Single-dose, Single-period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-Uproleselan Administered Via the Intravenous Route to Healthy Subjects (ADME Study of IV [14C]-Uproleselan in Healthy Subjects)
Brief Title: A Study in Healthy Volunteers to Investigate How Much Test Medicine [14C]-Uproleselan is Taken up by the Body When Administered Directly Into the Vein (IV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GMI-1271-104
Record Dates: First submitted 2018-07-23; First posted 2018-07-30 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — uproleselan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single IV administration of [14C]-Uproleselan (Experimental)
  Interventions: Drug: Uproleselan

INTERVENTIONS:
Drug: Uproleselan — [14C]-Uproleselan

SUMMARY:
The purpose of the study is to measure how the radiolabelled test medicine [14C]-Uproleselan (GMI-1271) is taken up, broken down and removed from the body when given intravenously (into a vein) in a group of 6 males. 'Radiolabelled' means that the test medicine has a radioactive component which helps us to track where the drug is in the body. Blood urine and fecal samples will be collected at specific times throughout the study to measure amounts of the test medicine in the body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age 30 to 65 years of age
* Body mass index (BMI) of 18.0 to 35.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
* Must be willing and able to communicate and participate in the whole study
* Must have regular bowel movements (ie, average stool production of ≥1 and ≤3 stools per day)
* Must provide written informed consent
* Must adhere to the contraception requirements

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the previous 3 months
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption
* Current smoking or use of tobacco products or substitutes.
* Current users of e-cigarettes and nicotine replacements products
* Radiation exposure
* Subjects who have completed 2 ADME studies in the last 12 months
* Clinically significant abnormal biochemistry, hematology or urinalysis
* Positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Evidence of renal impairment at screening
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug
* Vaccination with any live vaccine within 4 weeks of study drug administration

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Mass Balance Recovery | up to 8 days
  Urine and feces will be collected at different time points and the radioactivity will be measured. The recovery will be expressed as percentage of radioactivity administered
Tmax | up to 8 days
  The time from dosing at which Cmax was apparent
Cmax | up to 8 days
  maximum observed concentration
AUC(0-last) | up to 8 days
  area under the curve from 0 time to last measurable concentration
AUC(0-inf) | up to 8 days
  area under the curve from 0 time extrapolated to infinity
AUC%extrap | up to 8 days
  percentage of AUC(0-inf) extrapolated beyond last measured time point
lambda-z | up to 8 days
  the apparent elimination rate constant
T1/2 | up to 8 days
  the apparent elimination half-life
CI | up to 8 days
  clearance, the apparent volume cleared of parent drug per unit time after intravenous administration
Vx | up to 8 days
  the apparent volume of distribution after intravenous administration
MRT | up to 8 days
  mean residence time
Ae(urine) | up to 8 days
  the amount of Uproleselan excreted in the urine expressed as a percentage of the administered dose
%Ae(urine) | up to 8 days
  the amount of Uproleselan excreted in the urine expressed as a percentage of the administered dose
CLr | up to 8 days
  renal clearance: the apparent volume of plasma cleared of Uproleselan per unit time via renal elimination, calculated as: CLr = Ae (urine) / AUC

CONTACTS AND LOCATIONS:
Overall Officials: Nand Singh, MD,DPM,MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences Limited, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No